CLINICAL TRIAL: NCT02169063
Title: PET Imaging as a Biomarker of Systemic Treatment Response for Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Carbon-11 Acetate and Fluorine F 18 Sodium Fluoride PET as a Biomarker of Treatment Response in Patients With Hormone Resistant Metastatic Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8021; NCI-2014-01203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8021 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carbon-11 acetate; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (11C-acetate, 18F-fluoride, PET) (Experimental): Patients receive carbon-11 acetate IV and fluorine F 18 sodium fluoride IV over 1 minute and undergo PET at baseline and at 6-12 weeks after systemic therapy starts.
  Interventions: Radiation: carbon-11 acetate; Radiation: fluorine F 18 sodium fluoride; Procedure: positron emission tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: carbon-11 acetate — Given IV
Radiation: fluorine F 18 sodium fluoride — Given IV
  Other Names: 18 F-NaF; F-18 NaF
Procedure: positron emission tomography — Undergo 11C-acetate and 18F-fluoride PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies carbon-11 acetate and fluorine F 18 sodium fluoride positron emission tomography (PET) as a biomarker of treatment response in patients with prostate cancer that does not respond to treatment with hormones and has spread to other parts of the body. Carbon-11 acetate and fluorine F 18 sodium fluoride are radioactive drugs that may be useful in evaluating prostate cancer activity in response to treatment. Comparing results of diagnostic procedures such as carbon-11 acetate and fluorine F 18 sodium fluoride PET done before and after therapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate that carbon-11 acetate (11C-acetate) and 18F-fluoride (fluorine F 18 sodium fluoride) PET scans change as a result of treatment for men with metastatic castration-resistant prostate cancer by comparison of pre-treatment and 6-12 week post-treatment images (standardized uptake value [SUV], influx constant [Ki], and rate constant [K1]) with clinical response measures.

SECONDARY OBJECTIVES:

I. Compare results from 11C-acetate and 18F-fluoride PET scanning with the patient's clinical bone scan and determine which predicts clinical response better.

II. Compare changes in 11C-acetate and 18F-fluoride PET with changes in prostate-specific antigen (PSA) level.

III. Compare changes in 11C-acetate and 18F-fluoride PET with changes in urinary N-telopeptide and bone alkaline phosphatase.

IV. Determine if either baseline uptake or change in uptake for 11C-acetate and/or 18F-fluoride PET is correlated with progression-free survival by Prostate Cancer Working Group 2 (PCWG2) criteria (Scher, 2008).

V. Determine if either baseline uptake or change in uptake by 11C-acetate and/or 18F-fluoride PET is correlated with skeletal-related events (SREs) defined as radiographic pathologic fracture, need for radiation to bone, need for surgery, spinal cord compression or malignant hypercalcemia.

VI. Percentage of patients that experience adverse events by Common Terminology Criteria for Adverse Events, version 4.0.

VII. For patients who have tissue/blood biomarkers obtained for other indications, directly compare baseline uptake and change in uptake by 11C-acetate and/or 18F-fluoride PET with those biomarkers.

OUTLINE:

Patients receive carbon-11 acetate intravenously (IV) and fluorine F 18 sodium fluoride IV over 1 minute and undergo PET at baseline and at 6-12 weeks after systemic therapy starts.

After completion of treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients preparing to receive systemic therapy to treat metastatic castration-resistant prostate cancer
* At the time of enrollment, patients must demonstrate evidence of castration-resistant prostate cancer with a documented castrate level of serum total testosterone (< 50 ng/dL) while on continuous androgen deprivation therapy
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific screening procedures
* Be willing and able to comply with scheduled visits and other trial procedures
* Presence of at least one measurable or detectable metastasis as defined by bone scintigraphy, computed tomography (CT) scan appearance (magnetic resonance imaging [MRI] if indicated), or plain x-ray appearance

Exclusion Criteria:

* Any condition that would alter the patient's mental status, prohibiting the basic understanding and/or authorization of informed consent
* A serious underlying medical condition that would otherwise impair the patient's ability to receive treatment and imaging studies
* Expected lifespan of 12 weeks or less
* Extremely poor intravenous access, prohibiting the placement of a peripheral IV line for injection of radiotracer
* Radiation treatment to bone less than 4 weeks from the first PET scan
* Radiopharmaceutical treatment to bone less than 4 weeks from first PET scan
* Treatment with granulocyte-macrophage colony stimulating factor (GM-CSF) or granulocyte (G-CSF) within 4 weeks prior to first PET scan; patients should avoid treatment with these agents between the baseline and 6-12 treatment week imaging sessions
* Inability to lie still for imaging
* Weight > 300 pounds (lbs)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Changes in prostate cancer metastases as measured by 11C-acetate and 18F-fluoride PET in response to systemic therapy | Baseline to up to 12 weeks
  Percentage change between pre-treatment and post-therapy measurements will be computed for PET measures. Log transformations will be considered if the rates of change are highly skewed. Additionally, changes in PET measures will be analyzed descriptively by a stem-and-leaf plot.

SECONDARY OUTCOMES:
Clinical response data (response, stable disease or progression) | Up to 5 years
  Molecular imaging measures and clinical measures of treatment response, percentage change in PET derived imaging data will be compared to standard clinical parameters. Association between these two types of data decline will be analyzed using the mid-P adjustment to Fisher's exact test (Lancaster, 1961) to evaluate the potential clinical utility of change in 11C-acetate and 18F-fluoride as a biomarker for response.
Proportion of both 11C-acetate and 18F-fluoride PET scans and 99mTc bone scans in discovering suspicious sites that are later confirmed by standard bone scans | Up to 5 years
  Statistical significance of two proportions will be tested with a two-sample t-test for proportions (or nonparametric alternative).
Change in PSA parameters | Baseline to up to 30 days post-PET
  Spearman rank correlation will be used to examine correlations between PET parameters and continuous variable changes in PSA.
Change in urinary N-telopeptide | Baseline to up to 30 days post-PET
  Spearman rank correlation will be used to examine correlations between PET parameters and continuous variable changes in urinary N-telopeptide.
Change in bone alkaline phosphatase | Baseline to up to 30 days post-PET
  Spearman rank correlation will be used to examine correlations between PET parameters and continuous variable changes in bone alkaline phosphatase.
Progression-free survival (PFS) using PCWG2 | Up to 5 years
  Cox proportional hazards model will be used to investigate the predictive value of the differences in pre- and post- treatment measures on PCWG2 PFS.
SRE defined as radiographic pathologic fracture, need for radiation to bone, need for surgery, spinal cord compression or malignant hypercalcemia | Up to 5 years
  Cox proportional hazards model will be used to investigate the predictive value of the differences in pre- and post- treatment measures on time of first SRE.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Yu, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States